CLINICAL TRIAL: NCT02277626
Title: Comparison of the Airway Clearance Efficacy of Electro Flo 5000 and Vest Therapy in
Brief Title: Electro Flo 5000 and Vest Therapy
Acronym: EF/Vest
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Carlos Milla, Principal Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 24248
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2015-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Randomized Crossover to ElectroFlo (Experimental): Experimental: ElectroFlo 5000, then VEST Patients are randomized to a sequence of ElectroFlo 5000 on one visit and during the second visit, they cross-over to the Vest system.
  Interventions: Device: Electro Flo 5000
- Randomized Crossover to Vest (Experimental): Experimental: VEST, then ElectroFlo 5000 Patients are randomized to a sequence of Vest system on one visit and during the second visit, they cross-over to the ElectroFlo 5000.
  Interventions: Device: Incourage Vest System

INTERVENTIONS:
Device: Electro Flo 5000 — Airway clearance device
  Arms: Randomized Crossover to ElectroFlo
Device: Incourage Vest System — Airway Clearance Device
  Arms: Randomized Crossover to Vest

SUMMARY:
It is the goal of the proposed study to compare the efficacy, as assessed primarily by sputum weight, of these two different devices (the Electroflo 500 and VEST therapy) for airway clearance (AC) in CF patients with mild to moderate lung disease, who have stable lung health and perform AC at home as part of their routine therapeutic regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CF established by standard criteria (sweat chloride > 60 mmol/L and/or two alleles affected by gene mutations know to be associated with CF).
2. Age older than 12 years.
3. Known to consistently produce sputum.
4. Currently on a home therapeutic regimen that includes some form of AC performed at least 2 times daily.
5. FVC and FEV1 > 40%-predicted, and with stable lung function (no greater than a 10% variation in lung function parameters over the preceding 3 months).

Exclusion Criteria:

1. Hospitalization for CF pulmonary complications in the 2 months preceding enrollment.
2. Hemoptysis > 60 cc in a single episode in the 4 weeks preceding enrollment.
3. Chronic chest pain.
4. Participation in another interventional clinical trial in the previous 30 days. -

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Vest First Then ElectroFlo: Experimental: VEST, then ElectroFlo 5000 15 Patients were recruited from the Cystic Fibrosis Program at Stanford. All 15 patients were randomized to a sequence of Vest at one visit and during the second visit, they crossed-over to the ElectroFlo 5000.
  EnCourage Vest System: Airway Clearance Device
- ElectroFlo First Then Vest: Experimental: ElectroFlo 5000, then VEST 15 Patients were recruited from the Cystic Fibrosis Program at Stanford. All 15 patients were randomized to a sequence of ElectroFlo 5000 at one visit and during the second visit, they crossed-over to the Vest.
  Electro Flo 5000: Airway clearance device
Period: Overall Study
Arm/Group | Vest First Then ElectroFlo | ElectroFlo First Then Vest
Started | 6 | 9
Completed | 6 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Number of Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 33.33 [12.78 to 53.88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Wet Sputum Weight
Description: Sputum was collected in pre-measured cups in a blinded fashion
Time Frame: End of study visit per intervention
Measure: Mean (Full Range); unit: grams
Groups:
- Vest: VEST Arm
  Incourage Vest System: Airway Clearance Device
- Elecflo Arm: Elecflo Arm
  Electro Flo 5000: Airway clearance device
Arm/Group | Vest | Elecflo Arm
Number analyzed (Participants) | 15 | 15
grams | 3.8 [1.1 to 6.5] | 4.6 [0.8 to 8.4]

2. Secondary Outcome: Dry Sputum Weight
Description: Sputum was collected in pre-measured cups in a blinded fashion, dessicated and measured dry
Time Frame: End of study visit per intervention
Measure: Mean (Full Range); unit: gram
Groups:
- Vest Arm: Vest Arm
  Incourage Vest System: Airway Clearance Device
- ElectroFlo Arm: ElectroFlo Arm
  Electro Flo 5000: Airway clearance device
Arm/Group | Vest Arm | ElectroFlo Arm
Number analyzed (Participants) | 15 | 15
gram | 0.15 [0 to 0.31] | 0.18 [0 to 0.43]

3. Primary Outcome: Pulmonary Function Measured as a Percent Predicted BEFORE Therapy With Either ElectroFlo 5000 / VEST.
Description: Comparison of pulmonary function by doing spirometry testing on study patients during their Day 1 & Day 2 therapy sessions. Will also compare the results based on the therapies they receive.
Time Frame: End of study visit per intervention
Measure: Mean (Full Range); unit: percentage of predicted value
Arm/Group | ElectroFlo Arm | Vest Arm
Number analyzed (Participants) | 15 | 15
percentage of predicted value | 72.43 [55.81 to 89.05] | 72.93 [54.89 to 90.97]

4. Primary Outcome: Pulmonary Function Measured as a Percent Predicted AFTER Therapy With Either ElectroFlo 5000 / Vest.
Description: as for outcome 3
Time Frame: End of study visit per intervention
Measure: Mean (Full Range); unit: percentage of predicted value
Groups:
- Vest Arm: Vest Arm
  EnCourage Vest System: Airway Clearance Device
Arm/Group | Vest Arm | ElectroFlo Arm
Number analyzed (Participants) | 15 | 15
percentage of predicted value | 75.8 [57.36 to 94.24] | 75.73 [58.56 to 92.9]

5. Primary Outcome: Comfort Level After Receiving Therapy With Either ElectroFlo 5000 / Vest
Description: Comfort assessed on a scale of 1-10 by patients after therapy after each visit (1 being most comfortable, 10 being most un-comfortable)
Time Frame: End of study visit per intervention
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Vest Arm | ElectroFlo Arm
Number analyzed (Participants) | 15 | 15
units on a scale | 3.93 [0.84 to 7.02] | 2.67 [0.49 to 4.85]

ADVERSE EVENTS:
Arm/Group | Vest Arm | ElectroFlo Arm
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes